CLINICAL TRIAL: NCT05615090
Title: A Randomized Controlled Trials of Self-help Application for Eating Disorder Through Multifaceted Measurement
Brief Title: Self-help Application for Eating Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Eun Joo Kim, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3-2022-0342
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Eating Disorder in Adolescents and Young Adults

STUDY DESIGN:
Intervention Model Description: The waitlist group receives usual care for the first 8 weeks. After 8 weeks, the waitlist group begins the intervention and the immediate intervention group begins a maintenance phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Prepectoral) (Experimental): Participants received the Self-help app-based CBT-E for eating disorder for 8 weeks
  Interventions: Procedure: Arm I (Prepectoral),
- II (Subpectoral) (Other): Waiting list Wait-list control(participants will use the smartphone app after the intervention phase) The waitlist group will receive treatment as usual, Patients from the waitlist group will be offered access to App after a 8-weeks period.
  Interventions: Procedure: Arm II (Subpectoral)

INTERVENTIONS:
Procedure: Arm I (Prepectoral), — The intervention will be delivered through a smartphone app. The app provides users with ED symptom self-monitoring, psycho-education and relapse prevention in an evidence-based CBT-E.
  Arms: I (Prepectoral)
Procedure: Arm II (Subpectoral) — The intervention will be delivered through a smartphone app. The app provides users with ED symptom self-monitoring, psycho-education and relapse prevention in an evidence-based CBT-E.
  Arms: II (Subpectoral)

SUMMARY:
The purpose of this study is to determine whether mobile-based self-help CBT-E treatment for eating disorder can reduce eating disorder symptoms compared to the waitlist group

ELIGIBILITY:
Inclusion Criteria:

1. Aged 13-22 years
2. Owns a smartphone
3. Experienced at least one episode of binge eating over the past 4 weeks

Exclusion Criteria:

1. diagnosed with anorexia nervosa
2. BMI ≤ 17.5
3. having developmental disabilities, including autism, intellectual disabilities, schizophrenia, or other psychosis

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Cognitions assessed using EDE-Q global scores | Baseline, 8 weeks,16 weeks, 28 weeks
  The global score of Eating Disorder Examination Questionnaire (EDE-Q) has the 28-item scale of key attitudinal and behavioral ED symptoms. Higher scores indicate higher eating disorder symptomology.

SECONDARY OUTCOMES:
Change in concerns with body weight assessed using EDE-Q weight concern scores | Baseline, 8 weeks,16 weeks, 28 weeks
  EDE-Q subscales Higher scores indicate higher eating disorder symptomology.
Change in concerns with body shape assessed using EDE-Q shape concern scores | Baseline, 8 weeks,16 weeks, 28 weeks
  EDE-Q subscales Higher scores indicate higher eating disorder symptomology.
Change in restrained eating assessed using EDE-Q dietary restraint scores | Baseline, 8 weeks,16 weeks, 28 weeks
  EDE-Q subscales Higher scores indicate higher eating disorder symptomology.
Change in concerns with eating assessed using EDE-Q eating concern scores | Baseline, 8 weeks,16 weeks, 28 weeks
  EDE-Q subscales Higher scores indicate higher eating disorder symptomology.
Change in eating disorder symptoms assessed using the Eating Attitude Test | Baseline, 8 weeks,16 weeks, 28 weeks
  The Eating Attitude Test (EAT) is a 40-item, 6-point, self-report scale that measures dieting behaviors, food preoccupation, anorexia, bulimia, and concerns about being overweight. The total score (between 0 and 78) provides an overall risk score, where higher scores indicating greater risk of an eating disorder.
Change in addictive-like eating behaviors assessed using the Yale Food Addiction scale | Baseline, 8 weeks,16 weeks, 28 weeks
  The Yale Food Addiction Scale is a 35-item self-report inventory to identify people most likely to have an addiction to high-fat and/or high-sugar foods. The scale uses a combination of Likert and dichotomous scoring options. The YFAS provides two scoring options, a "symptom" count version that indicates the number of dependence symptoms experienced in the past 12 months and a "diagnostic" threshold that is met when three or more "symptoms" are present during the past 12 months and clinically significant impairment or distress is endorsed(Gearhardt et al., 2012).
Change in addictive-like eating behaviors assessed using the Yale Food Addiction Scale for Children | Baseline, 8 weeks,16 weeks, 28 weeks
  The Yale Food Addiction Scale for Children(YFAS-C) is a 25-item, 5-point self-report scale with higher scores indicating more food addiction symptoms in children. Items 1 to 18 are rated on a 5-point Likert scale and Items 19 to 25 are rated on a dichotomous (0 = no; 1 = yes) scale.
Change in emotion regulation problems assessed using the Difficulties in Emotion Regulation Scale | Baseline, 8 weeks,16 weeks, 28 weeks
  The Difficulties in Emotion Regulation Scale(DERS) is the 36 items self-report scale to asks respondents how they relate to their emotions. Scores are presented as a total score as well as a score for each of the 6 subscales. Higher scores mean greater problems with emotion regulation.
Change in Depression symptoms assessed using the Beck Depression Inventory | Baseline, 8 weeks,16 weeks, 28 weeks
  The Beck Depression Inventory (BDI) is a 21-item self-reporting questionnaire for assessing the severity of depression. The total score range from 0 to 63 and 0-9 indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression and 30-63: indicates severe depression.
Change in anxiety symptoms assessed using the State-Trait Anxiety Inventory | Baseline, 8 weeks,16 weeks, 28 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale. Higher scores indicate greater anxiety
Change in assessed the impact an eating disorder has on psychosocial functioning using The Clinical Impairment Assessment Questionnaire (CIA) | Baseline, 8 weeks,16 weeks, 28 weeks
  The Clinical Impairment Assessment questionnaire (CIA) is a 16-items self-report measure to assess psychosocial impairment resulting from eating disorder features. Possible scores range between 0 - 48, with higher scores indicating more impairment and lower scores indicating less impairment.
Change in self-esteem assessed using the Rosenberg self-esteem scale (RSES) | Baseline, 8 weeks,16 weeks, 28 weeks
  The Rosenberg Self-Esteem Scale(RSES) is a A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self. The total score is from 0 to 30, with higher scores representing higher self-esteem.
Change in the body attitudes associated with desiring a thinner assessed using the Eating Disorder Inventory-2, Drive for Thinness | Baseline, 8 weeks,16 weeks, 28 weeks
  Drive for thinness (DT), a subscale of the Eating Disorder Inventory (EDI), is a self-report measure of disordered eating attitudes about body image, weight, and shape. The total score is from 0 to 21. Higher scores mean an excessive concern with dieting, preoccupation with weight, and fear of weight gain
Change in eating disorder symptoms assessed using the Korean version of the Eating disorder Diagnostic Scale | Baseline, 8 weeks,16 weeks
  The Eating Disorder Diagnostic Scale (EDDS) is a 22-item self-report questionnaire designed to measure eating disorders symptomatology
Change in the heart rate variability | Baseline, 8 weeks,16 weeks
  The heart rate variabilities the physiological recordings of the variation in the time interval between consecutive heartbeats in milliseconds. This measures only those who want it
Change in brain activities recorded with functional near-infrared spectroscopy (fNIRS) | Baseline, 8 weeks
  Functional near-infrared spectroscopy (fNIRS) is a tool to measure functional brain activities using the changes of optical absorption in the brain through the intact skull. This tool measures only those who want it, and the target number of participants is 40.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Gearhardt AN, White MA, Masheb RM, Morgan PT, Crosby RD, Grilo CM. An examination of the food addiction construct in obese patients with binge eating disorder. Int J Eat Disord. 2012 Jul;45(5):657-63. doi: 10.1002/eat.20957. Epub 2011 Aug 30. PMID 22684991